CLINICAL TRIAL: NCT01261130
Title: Phase 1 Study of the Safety and Immunogenicity of Na-GST-1/Alhydrogel® With or Without GLA-AF in Brazilian Adults
Brief Title: Safety and Immunogenicity of a Human Hookworm Candidate Vaccine With or Without Additional Adjuvant in Brazilian Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Maria Elena Bottazzi PhD, Sponsor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SVI-10-01
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Hookworm Infection; Hookworm Disease
Keywords: Human Hookworm Vaccine Initiative; HHVI; Human Hookworm; Hookworm; Hookworm Disease; N. americanus; Soil-transmitted helminth infection; Intestinal blood loss; Iron deficiency anemia
MeSH Terms: conditions — Hookworm Infections; Ancylostomiasis; Anemia, Iron-Deficiency | interventions — D-Worm; Granuflex E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (13):
- Part I-A: 10μgNaGST1/Alhydrogel (Experimental): Part I (non-endemic area), Formulation A
  Interventions: Biological: 10 μg Na-GST-1/Alhydrogel
- Part I-B: 30μgNaGST1/Alhydrogel (Experimental): Part I (non-endemic area), Formulation B
  Interventions: Biological: 30 μg Na-GST-1/Alhydrogel
- Part I-C: 100μgNaGST1/Alhydrogel (Experimental): Part I (non-endemic area), Formulation C
  Interventions: Biological: 100 μg Na-GST-1/Alhydrogel
- Part I-D: 10μgNaGST1/Alhydrogel/GLA (Experimental): Part I (non-endemic area), Formulation D
  Interventions: Biological: 10 μg Na-GST-1/ Alhydrogel/GLA-AF
- Part I-E: 30μgNaGST1/Alhydrogel/GLA (Experimental): Part I (non-endemic area), Formulation E
  Interventions: Biological: 30 μg Na-GST-1/Alhydrogel/GLA-AF
- Part I-F: 100μgNaGST1/Alhydrogel/GLA (Experimental): Part I (non-endemic area), Formulation F
  Interventions: Biological: 100 μg Na-GST-1/Alhydrogel/GLA-AF
- Part II-A: 10μgNaGST1/Alhydrogel (Experimental): Part II (endemic area), Formulation A
  Interventions: Biological: 10 μg Na-GST-1/Alhydrogel
- Part II-B: 30μgNaGST1/Alhydrogel (Experimental): Part II (endemic area), Formulation B
  Interventions: Biological: 30 μg Na-GST-1/Alhydrogel
- Part II-C: 100μgNaGST1/Alhydrogel (Experimental): Part II (endemic), Formulation C
  Interventions: Biological: 100 μg Na-GST-1/Alhydrogel
- Part II-D: 10μgNaGST1/Alhydrogel/GLA (Experimental): Part II (endemic area), Formulation D
  Interventions: Biological: 10 μg Na-GST-1/ Alhydrogel/GLA-AF
- Part II-E: 30μgNaGST1/Alhydrogel/GLA (Experimental): Part II (endemic area), Formulation E
  Interventions: Biological: 30 μg Na-GST-1/Alhydrogel/GLA-AF
- Part II-F: 100μgNaGST1/Alhydrogel/GLA (Experimental): Part II (endemic area), Formulation F
  Interventions: Biological: 100 μg Na-GST-1/Alhydrogel/GLA-AF
- Part II-G: Butang® hepatitis B vaccine (Active Comparator): Part II (endemic), HepB comparator
  Interventions: Biological: Butang® hepatitis B vaccine

INTERVENTIONS:
Biological: 10 μg Na-GST-1/Alhydrogel — 3 doses 10 μg Na-GST-1/Alhydrogel administered at 56 day intervals
  Other Names: Formulation A
  Arms: Part I-A: 10μgNaGST1/Alhydrogel; Part II-A: 10μgNaGST1/Alhydrogel
Biological: 30 μg Na-GST-1/Alhydrogel — 3 doses 30 μg Na-GST-1/Alhydrogel administered at 56 day intervals
  Other Names: Formulation B
  Arms: Part I-B: 30μgNaGST1/Alhydrogel; Part II-B: 30μgNaGST1/Alhydrogel
Biological: 100 μg Na-GST-1/Alhydrogel — 3 doses 100 μg Na-GST-1/Alhydrogel administered at 56 day intervals
  Other Names: Formulation C
  Arms: Part I-C: 100μgNaGST1/Alhydrogel; Part II-C: 100μgNaGST1/Alhydrogel
Biological: 10 μg Na-GST-1/ Alhydrogel/GLA-AF — 3 doses 10 μg Na-GST-1/ Alhydrogel/GLA-AF administered at 56 day intervals
  Other Names: Formulation D
  Arms: Part I-D: 10μgNaGST1/Alhydrogel/GLA; Part II-D: 10μgNaGST1/Alhydrogel/GLA
Biological: 30 μg Na-GST-1/Alhydrogel/GLA-AF — 3 doses 30 μg Na-GST-1/Alhydrogel/GLA-AF administered at 56 day intervals
  Other Names: Formulation E
  Arms: Part I-E: 30μgNaGST1/Alhydrogel/GLA; Part II-E: 30μgNaGST1/Alhydrogel/GLA
Biological: 100 μg Na-GST-1/Alhydrogel/GLA-AF — 3 doses 100 μg Na-GST-1/Alhydrogel/GLA-AF administered at 56 day intervals
  Other Names: Formulation F
  Arms: Part I-F: 100μgNaGST1/Alhydrogel/GLA; Part II-F: 100μgNaGST1/Alhydrogel/GLA
Biological: Butang® hepatitis B vaccine — 3 doses Butang® hepatitis B vaccine administered at 56 day intervals
  Arms: Part II-G: Butang® hepatitis B vaccine

SUMMARY:
This two part study will evaluate the safety and immunogenicity of two formulations of Na-GST-1, first in hookworm-naïve individuals using an open-label design, and then in adults living in an area of endemic hookworm infection using a randomized, double-blind design. The two formulations to be evaluated are Na-GST-1 adsorbed to an adjuvant, Alhydrogel®, and Na-GST-1 adsorbed to Alhydrogel® and administered with GLA-AF.

DETAILED DESCRIPTION:
Human hookworm infection is a soil-transmitted helminth infection caused by the nematode parasites Necator americanus and Ancylostoma duodenale. It is one of the most common chronic infections of humans, afflicting up to 740 million people in the developing nations of the tropics. The largest number of cases occurs in impoverished rural areas of sub-Saharan Africa, Southeast Asia, China, and the tropical regions of the Americas. Approximately 3.2 billion people are at risk for hookworm infection in these areas. N. americanus is the most common hookworm worldwide, whereas A. duodenale is more geographically restricted.

The primary approach to hookworm control worldwide has been the frequent and periodic mass administration of benzimidazole anthelminthics to school-aged children living in high-prevalence areas. In 2001, the World Health Assembly adopted Resolution 54.19 which urges member states to provide regular anthelminthic treatment to high-risk groups with the target of regular treatment of at least 75% of all at-risk school-aged children. However, the cure rates for a single dose of a benzimidazole varies with rates as low as 61% (400 mg) and 67% (800 mg) for albendazole and 19% (single dose) and 45% (repeated dose) for mebendazole being reported. These concerns have prompted interest in developing alternative tools for hookworm control. Vaccination to prevent the anemia associated with moderate and heavy intensity hookworm infection would alleviate the public health deficiencies of drug treatment alone.

The current strategy for development of Human Hookworm candidate vaccines is focused on antigens expressed during the adult stage of the hookworm life cycle which play a role in digesting the host hemoglobin, used by the worm as an energy source. These antigens are relatively hidden from the human immune system during natural infection, and hence have a low likelihood of inducing antigen-specific IgE in exposed/infected individuals, reducing the potential for allergic reaction upon vaccination.

The nutritional and metabolic requirements of the adult hookworm living in the human intestine are dependent upon degradation of host hemoglobin that has been ingested by the worm. N. americanus hookworms depend on host hemoglobin for survival. Following hemolysis, adult hookworms use an ordered cascade of hemoglobinases to cleave hemoglobin into smaller molecules. Following hemoglobin digestion, the freed heme generates toxic oxygen radicals that can be bound and detoxified by molecules such as glutathione S-transferase-1 (GST-1). GST-1 of N. americanus (Na-GST-1) is a critical enzyme that plays a role in parasite blood feeding; when used as a vaccine, the investigators hypothesize that the antigen will induce anti-enzyme neutralizing antibodies that will interfere with parasite blood-feeding and cause parasite death or reduce worm fecundity.

Following its selection as a candidate antigen Na-GST-1 has been successfully manufactured and tested in the laboratory and in animals with both Alhydrogel® (aluminum hydroxide suspension)and Alhydrogel® plus Gluco-Pyranosylphospho-Lipid A Aqueous Formulation (GLA-AF). Na-GST-1 has been shown to be pure, potent, and stable when administered as either of these two formulations.

The Na-GST-1 vaccine formulations to be tested in this study consist of the 24 kDa recombinant protein Na-GST-1 adsorbed to Alhydrogel® either with or without the addition of GLA-AF. For the Na-GST-1/GLA-AF formulation, the GLA-AF will be added to the Alhydrogel® formulation immediately prior to immunization. The active ingredient in both vaccine formulations is the recombinant Na-GST-1 protein that is derived by fermentation of Pichia pastoris yeast cells genetically engineered to express Na-GST-1.

In this first-in-human study, the evaluation of the safety and immunogenicity of the Na-GST-1 and Na-GST-1/GLA-AF formulations will be conducted in two parts. First, healthy adults who have not been infected with or exposed to hookworm will be enrolled in the urban center of Belo Horizonte, Brazil. Hookworm in Brazil is primarily a rural disease and is uncommon in developed urban areas such as Belo Horizonte. If no significant safety concerns are observed in these volunteers, the study will proceed to enroll and vaccinate healthy adults in a hookworm-endemic region of the state of Minas Gerais, Brazil. The vaccine formulations will be tested in both populations (i.e., non-endemic and endemic areas), given the possibility that the safety profile of the vaccine formulations may be different in a population that has been chronically exposed to the antigen contained in these vaccines.

In Part I of the study, 36 volunteers will be enrolled into one of six cohorts. In the first cohort, 6 individuals will receive the 10 µg dose of Na-GST-1/Alhydrogel®; in the second cohort, 6 individuals will receive the 10 µg dose of Na-GST-1/Alhydrogel®/GLA-AF; in the third and fourth cohorts, 6 volunteers each will receive 30 µg Na-GST-1/Alhydrogel® and Na-GST-1/Alhydrogel®/GLA-AF, respectively; while in the fifth and sixth cohorts, 6 volunteers each will receive 100 µg Na-GST-1/Alhydrogel® and Na-GST-1/Alhydrogel®/GLA-AF, respectively. Enrollment of these cohorts will be staggered by one-week intervals: Cohorts 2 and 3 will be enrolled and begin vaccinations 1 week after Cohort 1, Cohorts 4 and 5 will be vaccinated 1 week after Cohorts 2 and 3, and Cohort 6 will be vaccinated 1 week after Cohorts 4 and 5.

In Part II of the study, 66 volunteers will be progressively enrolled into one of six dose cohorts. In the first, third and fifth cohorts, volunteers will be randomized to receive either Na-GST-1/Alhydrogel® (n=8) or Butang® (n=2), while in the second, fourth and sixth cohorts, volunteers will be randomized to receive either Na-GST-1/Alhydrogel® (n=2) or Na-GST-1/Alhydrogel®/GLA-AF (n=10). Volunteers randomized to receive Na-GST-1 will receive either the 10 µg, 30 µg or 100 µg dose. In order to ensure that the vaccine formulations will be evaluated in individuals recently infected with hookworm, at least 4 individuals will be enrolled into each of the Part II chohorts who were infected with hookworm based on the fecal exam conducted during the screening for the study, or who had a documented infection within 3 months of the date planned for the first vaccination for the participant.

The investigators have chosen the Butang® hepatitis B vaccine (Instituto Butantan, Sao Paulo, Brazil) as the comparator vaccine for five principal reasons: (1) it is likely to confer some benefit to the participants receiving it, (2) it has an established safety record, (3) it is a yeast-derived recombinant protein adsorbed to an aluminum-containing immunostimulant, (4) it has the same physical appearance as Na-GST-1 immunostimulanted with Alhydrogel, and (5) its dosing schedule permits easy incorporation into the study design. Furthermore, Butang® is the most widely-used hepatitis B vaccine in Brazil, with over 15 million doses distributed annually.

Each participant will recieve 3 doses of the assigned study agent given in 56 day intervals (i.e. Day 0, Day 56 and Day 112). The trial is expected to last for a total of 24 months. Each participant will be followed for 16 months from the time of the first injection.

Safety parameters will be monitored throughout both parts of the study. The primary immunological endpoint for both parts will be the measurement of the antigen-specific antibody response.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 45 years, inclusive.
* Good general health as determined by means of the screening procedure.
* Available for the duration of the trial (42 weeks).
* Willingness to participate in the study as evidenced by signing the informed consent document.
* If found to be infected with hookworm during screening, has completed a course of three doses of albendazole.

Exclusion Criteria:

* Pregnancy as determined by a positive urine β-hCG (if female).
* Participant unwilling to use reliable contraception methods up until one month following the third immunization (if female).
* Currently lactating and breast-feeding (if female).
* Inability to correctly answer all questions on the informed consent comprehension questionnaire.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, diabetes, or renal disease by history, physical examination, and/or laboratory studies.
* Known or suspected immunodeficiency.
* Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 1.25-times the upper reference limit).
* Laboratory evidence of renal disease (serum creatinine greater than 1.25-times the upper reference limit, or more than trace protein or blood on urine dipstick testing).
* Laboratory evidence of hematologic disease (absolute leukocyte count <3000/mm3 or >12.5 x 103/mm3; hemoglobin <10.3 g/dl or <11.0 g/dl [females in Americaninhas and Belo Horizonte, respectively] or <11.0 g/dl or <12.0 [males in Americaninhas and Belo Horizonte, respectively); absolute lymphocyte count <900/mm3; or platelet count <120,000/mm3).
* Laboratory evidence of a coagulopathy (PTT or PT INR greater than 1.1-times the upper reference limit [in Belo Horizonte] or PT INR greater than 1.3 [Americaninhas]).
* Serum glucose (random) greater than 1.2-times the upper reference limit.
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
* Participation in another investigational vaccine or drug trial within 30 days of starting this study.
* Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma as defined by the need for regular use of inhalers or emergency clinic visit or hospitalization within the last 6 months.
* Positive ELISA for HCV.
* Positive ELISA for HBsAg.
* Positive ELISA for HIV.
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study.
* Receipt of a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to entry into the study.
* History of a surgical splenectomy.
* Receipt of blood products within the past 6 months.
* History of allergy to yeast.
* Anti-Na-GST-1 IgE antibody level above 0.35 kUA/L by the ImmunoCAP method.
* For Part I only: history of previous infection with hookworm; residence for more than 6 months in a hookworm-endemic area; or, positive for hookworm infection on screening microscopic fecal examination.
* For Part II only: previous receipt of a primary series of any hepatitis B vaccine.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2011-11; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Immediate vaccine related adverse events | 2 hours post vaccination
  Frequency of vaccine-related AEs, graded by severity, for each dose and formulation of Na-GST-1

SECONDARY OUTCOMES:
IgG antibody response to Na-GST-1 | 126 days post dose 1
  Dose and formulation of Na-GST-1 that generates the highest IgG antibody response at Day 126, as determined by an indirect enzyme-linked immunosorbent assay (ELISA)
Duration of antibody response to Na-GST-1 | 290 days post dose 1
  Duration of anti-GST-1 antibody, up to Day 290, as determined by an indirect enzyme-linked immunosorbent assay (ELISA)
Exploratory cellular immune response to Na-GST-1 | Up to 290 days post dose 1
  Cellular immune responses to the Na-GST-1 antigen both before and after immunization

CONTACTS AND LOCATIONS:
Overall Officials: David Diemert, MD, Principal Investigator — Albert B. Sabin Vaccine Institute
Locations (2):
- Brazil (2):
  - Americaninhas Vaccine Center, Americaninha, Minas Gerais
  - Centro de Pesquisas René Rachou - FIOCRUZ, Belo Horizonte, Minas Gerais

REFERENCES:
- [Derived] Diemert DJ, Freire J, Valente V, Fraga CG, Talles F, Grahek S, Campbell D, Jariwala A, Periago MV, Enk M, Gazzinelli MF, Bottazzi ME, Hamilton R, Brelsford J, Yakovleva A, Li G, Peng J, Correa-Oliveira R, Hotez P, Bethony J. Safety and immunogenicity of the Na-GST-1 hookworm vaccine in Brazilian and American adults. PLoS Negl Trop Dis. 2017 May 2;11(5):e0005574. doi: 10.1371/journal.pntd.0005574. eCollection 2017 May. PMID 28464026